CLINICAL TRIAL: NCT06895772
Title: Analysis of Microbial Community Characteristics in Intestinal Mucosal Tissue of Patients With Crohn's Disease
Brief Title: Microbial Community Characteristics in Intestinal Mucosal Tissue of Patients With CD
Status: Active, not recruiting | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Gastroenterology Department, Qilu Hospital of Shandong University
Other Study IDs: 2025-SDU-Qilu-01
Record Dates: First submitted 2025-03-10; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Crohn's Disease (CD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD patients: Before receiving treatment, 2-4 biopsy samples of small or large intestinal mucosa are collected from Crohn's disease patients, including both lesional and normal tissues.
  During follow-up endoscopy performed 3-12 months after treatment for Crohn's disease patients, either due to symptoms or routine re-examination, 2-4 pieces of small or large intestinal mucosa are collected, including both lesional and normal tissues.
  Place the samples in a -80°C freezer for storage and submit them for 5R 16S high-throughput sequencing.
- Healthy individuals: Collect 1-2 pieces of large or small intestinal mucosa from healthy individuals with no symptoms who undergo colonoscopy and show no lesions, or from patients who undergo small intestinal endoscopy due to symptoms but have negative examination results.
  Place the samples in a -80°C freezer for storage and submit them for 5R 16S high-throughput sequencing.

SUMMARY:
The characteristics of the intestinal microbiota in Crohn's disease and their relationship with disease pathogenesis have not yet been fully elucidated. Therefore, this study aims to analyze the microbial community characteristics in the intestinal mucosal tissue of Crohn's disease patients and fill this knowledge gap. Additionally, this research holds significant importance for understanding the etiology of Crohn's disease and predicting treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease undergoing endoscopic examination
* Healthy individuals with no symptoms undergoing colonoscopy without any lesions detected
* Patients undergoing small intestinal endoscopy due to symptoms but with negative examination results.
* Age between 18 and 80 years.
* Patients or authorized family members sign the relevant informed consent forms.

Exclusion Criteria:

* Patients with concurrent digestive system diseases that may affect the study results, including tumors, infections, or other autoimmune diseases.
* Patients with concurrent non-digestive system diseases that may affect the study results, including tumors, infections, or autoimmune diseases.
* Patients who have taken probiotics or antibiotics within the past week.
* Patients with psychiatric disorders or other conditions that prevent them from cooperating with the study.
* Patients participating in other clinical trials that may interfere with the results of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CD patients or healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The characteristics of the intestinal microbiota in Crohn's disease | 12 months
  Analyze the characteristics of the microbiota within the intestinal mucosal tissue of patients with Crohn's disease；Analyze the differences in the microbiota between the lesional and normal intestinal mucosal tissues of patients with Crohn's disease；Analyze the differences in the microbiota within the intestinal mucosal tissue of patients with Crohn's disease before and after treatment.

SECONDARY OUTCOMES:
Contrast the characteristics of the intestinal microbiota in Crohn's disease and healthy individuals | 12 months
  Compare the differences in the microbiota within the intestinal mucosal tissue between patients with Crohn's disease and healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, doctor, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No